CLINICAL TRIAL: NCT02741557
Title: An Open-label, Randomized, Two-way Crossover, Single Dose, Pivotal Bioequivalence Study of a Fixed-dose Combination of Dolutegravir and Rilpivirine in Healthy Volunteers
Brief Title: Bioequivalence Study of a Fixed-dose Combination (FDC) of Dolutegravir (DTG) and Rilpivirine (RPV)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201676
Record Dates: First submitted 2016-04-14; First posted 2016-04-18 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-06

CONDITIONS: Infection, Human Immunodeficiency Virus; HIV Infections
Keywords: Fixed-dose Combination (FDC); Bioequivalence; Dolutegravir; Rilpivirine
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DTG/RPV FDC-DTG plus RPV (Experimental): Subjects will receive a single oral dose of DTG/RPV 50 mg/25 mg FDC tablet in Period 1 under fed state. After a washout period of at least 21 days, subjects will receive a single oral dose of separate tablet formulations of DTG 50 mg and RPV 25 mg together in Period 2 under fed state.
  Interventions: Drug: DTG; Drug: RPV; Drug: DTG/RPV FDC
- DTG plus RPV-DTG/RPV FDC (Experimental): Subjects will receive a single oral dose of separate tablet formulations of DTG 50 mg and RPV 25 mg together in Period 1 under fed state. After a washout period of at least 21 days, subjects will receive a single oral dose of DTG/RPV 50 mg/25 mg FDC tablet in Period 2 under fed state.
  Interventions: Drug: DTG; Drug: RPV; Drug: DTG/RPV FDC

INTERVENTIONS:
Drug: DTG — DTG is provided as a white, film-coated, round tablet containing DTG 50 mg, debossed with SV 572 on one side and 50 on the other side. Subjects will receive a single oral dose of DTG 50 mg tablet with 240 mL of water.
Drug: RPV — RPV is provided as a white to off-white, film-coated, round, biconvex tablet containing RPV 25 mg, debossed with TMC on one side and 25 on the other side. Subjects will receive a single oral dose of RPV 25 mg tablet with 240 mL of water.
Drug: DTG/RPV FDC — DTG/RPV FDC is provided as a pink, film coated, oval biconvex tablet containing FDC of DTG 50 mg and RPV 25 mg, debossed with SV J3T on one face. Subjects will receive a single oral dose of DTG/RPV 50 mg/25 mg FDC tablet with 240 mL of water.

SUMMARY:
The purpose of the study is to evaluate the bioequivalence between Fixed-dose Combination (FDC) tablet formulation of Dolutegravir (DTG) 50 milligrams (mg) and Rilpivirine (RPV) 25 mg versus co-administration of the separate tablet formulations of DTG 50 mg plus RPV 25 mg, in the fed state. This pivotal bioequivalence study, is to serve as a pharmacokinetic (PK) bridge to the ongoing Phase 3 trials with the separate agents. This study will be conducted under fed conditions to appropriately mimic the conditions in the Phase 3 trials. This is a single-center, randomized, open-label, 2-period, single-dose, crossover study. A minimum of 86 healthy adult subjects will be randomized such that a minimum of approximately 82 evaluable subjects complete the study. The total duration of participation of a subject in this study will be approximately 8 weeks which includes a screening visit within 30 days prior to the first dose of study drug, two treatment periods each with a single dose of study drug and a follow-up visit within 12-17 days after the last dose of study drug. There will be a washout of at least 21 days between each dose of study drug.

A blinded (for treatment) review of DTG and RPV plasma concentration data for approximately the first 40 subjects will be conducted. If the within-subject coefficients of variation (CVw%) for either DTG or RPV maximal drug concentration (Cmax) values are >=31%; a sample size re-estimation will be employed and additional subjects (beyond the 86 planned) will be randomized for treatment in the study. Following the re-estimation, it is possible that up to approximately 154 healthy adult subjects (68 new subjects in addition to the planned 86 subjects above) will be randomized such that a maximum of approximately 146 evaluable subjects could complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Age: Between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac evaluation (history, ECG).
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor if required agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=50 kilograms (kg) (110 pounds [lbs]) for men and >=45 kg (99 lbs) for women and body mass index (BMI) within the range 18.5-31.0 kg/square meter (m^2) (inclusive)
* Male or Female.

Females: A female subject is eligible to participate if she is not pregnant (as confirmed by a negative [serum or urine according to site standard procedure] human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies:

* Non-reproductive potential defined as: Pre-menopausal females with one of the following: Documented tubal ligation; Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion; Hysterectomy; Documented Bilateral Oophorectomy. Postmenopausal defined as 12 months of spontaneous amenorrhea. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment.
* Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study medication and until (at least five terminal half-lives OR until any continuing pharmacologic effect has ended, whichever is longer) after the last dose of study medication and completion of the follow-up visit.

  * Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the consent form and in the protocol.

Exclusion Criteria:

* ALT and bilirubin >1.5xupper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GlaxoSmithKline (GSK) Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 grams (g) of alcohol: 12 ounces (360 milliliters [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Positive results for drugs of abuse.
* Cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 30 days prior to screening.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood product in excess of 500 mL within 56 days.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination): Heart rate <45 and >100 beats per minute (bpm) for males and <50 and >100 bpm for females; PR Interval <120 and >220 milliseconds (msec); QRS Interval: <70 and >120 msec; and corrected QT (QTc) interval (Fridericia's) >450 msec.

Evidence of previous myocardial infarction (Does not include ST segment changes associated with repolarization).

* Any conduction abnormality (including but not specific to left or right complete bundle branch block, atrioventricular [AV] block [2nd degree or higher], Wolff-Parkinson-White [WPW] syndrome).
* Sinus Pauses > 3 seconds.
* Any significant arrhythmia which, in the opinion of the principal investigator or ViiV Healthcare (ViiV)/GSK medical monitor, will interfere with the safety for the individual subject.
* Non-sustained or sustained ventricular tachycardia (>=3 consecutive ventricular ectopic beats).

  * Employment with Janssen, ViiV, GSK, or with the Investigator or study site, with direct involvement in the proposed study or other studies under the direction of that Investigator or study site, as well as family members of the employees or the Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2016-10-24 (Actual); Study Completion 2016-10-24 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC) from time 0 extrapolated to infinity (AUC[0-inf]) of DTG and RPV in plasma | Blood samples will be collected at pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, 120, 168, 216, and 264 hours post-dose during the 2 treatment periods.
AUC from time 0 to the last measurable timepoint (AUC[0-t]) of DTG and RPV in plasma | Blood samples will be collected at pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, 120, 168, 216, and 264 hours post-dose during the 2 treatment periods.
Maximal drug concentration (Cmax) of DTG and RPV in plasma | Blood samples will be collected at pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, 120, 168, 216, and 264 hours post-dose during the 2 treatment periods.

SECONDARY OUTCOMES:
Absorption lag time (tlag) of DTG and RPV in plasma | Blood samples will be collected at pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, 120, 168, 216, and 264 hours post-dose during the 2 treatment periods.
Time to observed maximal drug concentration (tmax) of DTG and RPV in plasma | Blood samples will be collected at pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, 120, 168, 216, and 264 hours post-dose during the 2 treatment periods.
Time of last quantifiable concentration (t) of DTG and RPV in plasma | Blood samples will be collected at pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, 120, 168, 216, and 264 hours post-dose during the 2 treatment periods.
Half-life (t1/2) of DTG and RPV in plasma | Blood samples will be collected at pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, 120, 168, 216, and 264 hours post-dose during the 2 treatment periods.
Apparent terminal elimination phase rate constant (lambda z) of DTG and RPV in plasma | Blood samples will be collected at pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, 120, 168, 216, and 264 hours post-dose during the 2 treatment periods.
Percentage of AUC(0-inf) resulting from extrapolation (%AUCex) of DTG and RPV in plasma | Blood samples will be collected at pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, 120, 168, 216, and 264 hours post-dose during the 2 treatment periods.
AUC from time 0 to 24 hours (AUC[0-24]) of DTG and RPV in plasma | Blood samples will be collected at pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, 120, 168, 216, and 264 hours post-dose during the 2 treatment periods.
Apparent oral clearance (CL/F) of DTG and RPV in plasma | Blood samples will be collected at pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, 120, 168, 216, and 264 hours post-dose during the 2 treatment periods.
Apparent oral volume of distribution (Vz/F) of DTG and RPV in plasma | Blood samples will be collected at pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, 120, 168, 216, and 264 hours post-dose during the 2 treatment periods.
Last quantifiable concentration (Ct) of DTG and RPV in plasma | Blood samples will be collected at pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, 120, 168, 216, and 264 hours post-dose during the 2 treatment periods.
Concentration at 24 hours post-dose (C24) of DTG and RPV in plasma | Blood samples will be collected at pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 16, 24, 48, 72, 120, 168, 216, and 264 hours post-dose during the 2 treatment periods.
Change from baseline in 12-lead electrocardiogram (ECG) | Baseline and up to 8 weeks
Change from baseline in blood pressure (BP) | Baseline and up to 8 weeks
Change from baseline in heart rate (HR) | Baseline and up to 8 weeks
Number of subjects with any adverse events (AEs) and any serious adverse events (SAEs) | Up to 4 weeks
  An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, is associated with liver injury and impaired liver function.
Number of subjects with Grade 3/4 hematology parameters | Up to 8 weeks
Number of subjects with Grade 3/4 clinical chemistry parameters | Up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- [Background] Mehta R, Wolstenholme A, Di Lullo K, Fu C, Joshi S, Crauwels H, Givens N, Vanveggel S, Wynne B, Adkison K. Bioequivalence of a Fixed-Dose Combination Tablet of the Complete Two-Drug Regimen of Dolutegravir and Rilpivirine for Treatment of HIV-1 Infection. Antimicrob Agents Chemother. 2018 Aug 27;62(9):e00748-18. doi: 10.1128/AAC.00748-18. Print 2018 Sep. PMID 29987139